CLINICAL TRIAL: NCT03202797
Title: Optimizing Regulation of a Cochlear Implant in Patients With Functional Contralateral Audition Using an Evolutionary Algorithm.
Brief Title: Optimizing Regulation of a Cochlear Implant in Patients With Functional Contralateral Audition.
Acronym: BIMODALITE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Bozorg-SAADOUN 2016
Record Dates: First submitted 2017-06-21; First posted 2017-06-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Functional Contralateral Audition; Cochlear Implant
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: audiometric tests; Other: Questionnaires; Other: Settings of cochlear implants

INTERVENTIONS:
Other: audiometric tests — tone and speech audiometry
Other: Questionnaires — APHAB (Abbreviate Profile of Hearing Aid Benefit), HISQUI (Hearing Implant Sound Quality Index), Munich music questionnaire
Other: Settings of cochlear implants — pitch matching, evolutionary algorithm setting

SUMMARY:
360 million people in the world suffer from debilitating hearing deficiency. The cochlear implant is indicated in certain patients with severe profound deafness. The principle of the cochlear implant is to directly stimulate auditory nerve fibres by electrodes inserted in the cochlea. The steps in auditory rehabilitation are the surgical insertion of the cochlear implant, activation, and follow-up regulation. There is no formal consensus to define the exact modalities for regulation during activation or follow-up, but the principles are respected according to centres that regulate cochlear implant. Bimodal audition is the fact of having a cochlear implant and a contralateral hearing aid. In patients with cochlear implants, having binaural bimodal audition improves their auditory vocal performance in silence and in noisy environments. It needs to be considered when a second cochlear implant is not indicated for the contralateral ear. It has been shown that by allocating frequencies different from the default frequencies attributed by the manufacturer, intelligibility and perception of music are modified. The investigators therefore with to study this working hypothesis and to develop a simple protocol for the reallocation of frequencies in order to optimise auditory performance in the everyday lives of patients with implants by using an evolutionary algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided consent
* Patients over 18 years old
* Profound post-lingual deafness with a cochlear implant and a functional contralateral ear (normal audition or mild to severe deafness but with a hearing aid).
* Patients fitted with one of the following cochlear implants with the most recent processor: Cochlear, Med-El, Neurelec Oticon or Advanced Bionics.
* Patients with at least 6 months experience with the cochlear implant and using both aids for at least 6 hours per day.

Exclusion Criteria:

* Persons without health insurance cover
* Adults under guardianship
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Functional Contralateral Audition with Cochlear Implant
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Compare the audiometric test performances (tone and speech audiometry) before and after the cochlear implant settings based on the evolutionary algorithm with a signal to noise ratio of +5dB | Baseline and 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Saadoun A, Schein A, Pean V, Legrand P, Aho Glele LS, Bozorg Grayeli A. Frequency Fitting Optimization Using Evolutionary Algorithm in Cochlear Implant Users with Bimodal Binaural Hearing. Brain Sci. 2022 Feb 11;12(2):253. doi: 10.3390/brainsci12020253. PMID 35204015